CLINICAL TRIAL: NCT02424006
Title: A Prospective, Randomized, Open Label Clinical Trial to Evaluate the Safety and Effectiveness of the RHCIII-MPC Biosynthetic Cornea Compared to Human Cornea in Patients Requiring Anterior Lamellar Keratoplasty
Brief Title: Safety and Effectiveness of the RHCIII-MPC Biosynthetic Cornea in Patients Requiring Anterior Lamellar Keratoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L.V. Prasad Eye Institute (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Virender S Sangwan, MBBS, MS, Director, Center for Ocular Regeneration, L.V. Prasad Eye Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201503-001; LVPEI-RHCIII-MPC CORNEA (Other: Clinical Trial Registry - India)
Record Dates: First submitted 2015-04-10; First posted 2015-04-22 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2015-04

CONDITIONS: Leukoma
Keywords: keratoplasty; bioengineered cornea; donor cornea
MeSH Terms: conditions — Corneal Opacity

STUDY DESIGN:
Intervention Model Description: RHCIII-MPC Biosynthetic Cornea
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RHCIII-MPC cornea (Experimental): Patients of this arm will undergo RHCIII-MPC bioengineered cornea transplantation using anterior lamellar keratoplasty technique
  Interventions: Device: RHCIII-MPC cornea
- Donor cornea (Active Comparator): Patients of this arm will undergo human donor cornea transplantation using anterior lamellar keratoplasty technique
  Interventions: Device: Donor cornea

INTERVENTIONS:
Device: RHCIII-MPC cornea — Patients will undergo surgery using conventional anterior lamellar keratoplasty technique: diseased cornea will be trephined to 350 um of corneal thickness and then a lamellar dissection will be created. Trephine diameter will be 7.5 mm. Alternatively a femtosecond laser may be used to create the dissection. A RHCIII-MPC cornea 350 um thick and equal or 0.25 mm larger diameter is placed and sutured. The sutures are superimposed and the implant and the sutures covered with a bandage contact lens. The sutures and bandage lens will be removed later after the initial healing period of 4 weeks or as determined by physician depending on the implant epithelial coverage.
  Arms: RHCIII-MPC cornea
Device: Donor cornea — Patients will undergo surgery using conventional anterior lamellar keratoplasty technique: diseased cornea will be trephined to 350 um of corneal thickness and then a lamellar dissection will be created. Trephine diameter will be 7.5 mm. Alternatively a femtosecond laser may be used to create the dissection. A human donor cornea graft 350 um thick and 0.25 mm larger diameter is placed and sutured. The sutures will be removed in 3-6 months or as determined by physician.
  Arms: Donor cornea

SUMMARY:
In this study safety and effectiveness of bioengineered cornea comprising of interpenetrating networks of recombinant human type III collagen and synthetic phospholipid - phosphorylcholine - will be tested in patients with corneal scars (leukomas) after infection, trauma or keratoconus. Control group will consist of patients with the same condition who will undergo corneal transplantation - current standard of care.

DETAILED DESCRIPTION:
Recently developed and passed extensive pre-clinical testing collagen-phosphorylcholine(RHCIII-MPC) corneal substitute will be implanted in patient's corneas with corneal scar (leukoma) developed after infection, trauma or keratoconus using anterior lamellar keratoplasty technique, i.e. once patient's diseased anterior part of cornea is removed, either manually or with assistance of femtosecond laser, it will be substituted with proposed transparent implant. Control patients with same condition will be grafted with human donor cornea using the same surgical technique.

The investigators will test the safety and the effectiveness of developed biosynthetic corneas. Overall 20 patients are planned to recruit. They will be randomized in two groups - 10 patients will undergo RHCIII-MPC cornea implantation, another 10 will be impanted with human donor cornea. The patients will be follow-uped for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must sign and be given a copy of the written Informed Consent form.
* Subjects with best corrected distance visual acuity +1.0 LogMAR or worse as a result of corneal scar due to infection, injury or keratoconus in the operative eye.
* Subjects must be willing and able to return for scheduled follow-up examinations for 12 months after surgery.

Exclusion Criteria:

* Subjects with severe or life-threatening systemic disease.
* Subjects with uncontrolled hypertension.
* Subjects with uncontrolled diabetes or insulin-dependent diabetes.
* Subjects with glaucoma in either eye.
* Subjects with marked microphthalmos or aniridia in either eye.
* Subjects with any other serious ocular pathology, serious ocular complications at the time of surgery underlying serious medical conditions, based on the investigator's medical judgment.
* Subjects which are or lactating or who plan to become pregnant over the course of the clinical investigation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Safety (Degree of eye inflammation) | 12 months
  Degree of eye inflammation based on conjunctival injection, perifocal corneal haze, aqueous humor transparency, increased intraocular pressure and self reported postoperative pain. Each item is scored 0-4: 0 = no symptom, 4 = severe symptom.

SECONDARY OUTCOMES:
Biocompatability, degree of haze and/or vascularisation measured on a scale 0-4 | 12 months
  The implant/donor cornea graft biocompatability will be checked by degree of haze and/or vascularisation measured on a scale 0-4 (0 - transparent implant/graft, no vessels, 4 - haze does not allow visualizing pupil, vessels enter entire surface of implant/graft)
Visual acuity measured by LogMAR | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Virender S Sangwan, MBBS, MS, Principal Investigator — LV Prasad Eye Institute
Locations (1):
- L V Prasad Eye Institute, Centre for Ocular Regeneration, Hyderabad, India

REFERENCES:
- [Result] Liu W, Deng C, McLaughlin CR, Fagerholm P, Lagali NS, Heyne B, Scaiano JC, Watsky MA, Kato Y, Munger R, Shinozaki N, Li F, Griffith M. Collagen-phosphorylcholine interpenetrating network hydrogels as corneal substitutes. Biomaterials. 2009 Mar;30(8):1551-9. doi: 10.1016/j.biomaterials.2008.11.022. Epub 2008 Dec 20. PMID 19097643
- [Result] Fagerholm P, Lagali NS, Ong JA, Merrett K, Jackson WB, Polarek JW, Suuronen EJ, Liu Y, Brunette I, Griffith M. Stable corneal regeneration four years after implantation of a cell-free recombinant human collagen scaffold. Biomaterials. 2014 Mar;35(8):2420-7. doi: 10.1016/j.biomaterials.2013.11.079. Epub 2013 Dec 25. PMID 24374070